CLINICAL TRIAL: NCT02452021
Title: An Observational Study of Pencil Beam Scanning (PBS) Proton Radiotherapy (RT) as a Component of Trimodality Therapy for Esophageal Cancer
Brief Title: Pencil Beam Scanning Proton Radiotherapy for Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Christopher (Chris) L. Hallemeier, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 15-002155
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study designed to observe the toxicity and efficacy of PBS proton RT for patients with esophageal cancer undergoing trimodality therapy. The investigators hypothesize that PBS proton RT will be associated with a favorable adverse event profile and quality of life, with similar disease control outcomes, relative to historical comparisons of patients treated with photon RT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histological confirmation of adenocarcinoma or squamous cell carcinoma of the esophagus (mid, distal, or GE junction)
* Stage T1N1-3M0 or T2-4N0-3M0 by American Joint Commission on Cancer (AJCC) 7th edition
* Tumor extends ≤ 5 cm into gastric cardia, based on EGD and PET/CT
* ECOG Performance Status (PS) 0-2 (Appendix I)
* Surgical consultation to confirm that patient is an appropriate candidate for esophagectomy
* Medical oncology consultation to confirm that patient is an appropriate candidate for chemotherapy
* Planned to receive standard of care neoadjuvant CRT, consisting of PBS proton RT (50 Gy/25 fractions) and concurrent chemotherapy (weekly carboplatin and paclitaxel), followed by surgical resection
* Ability to complete questionnaire(s) by themselves or with assistance.
* Provide informed written consent.
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

Note: During the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up.

* Willing to sign consent onto the Mayo Clinic Radiotherapy Patient Outcomes Registry and Biobanking study, IRB number 15-000136

Exclusion Criteria:

* Cervical or upper esophageal tumors with any part of tumor < 24 cm from incisors
* Prior chemotherapy or RT for esophageal cancer
* History of RT to the thorax
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of adverse events.
* Immunocompromised patients and patients known to be HIV positive and not currently receiving antiretroviral therapy. NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any investigational agent which would be considered as a treatment for the primary neoplasm.
* Other active malignancy ≤ 1 year prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer.
* History of myocardial infarction ≤6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with non-metastatic esophageal cancer who are candidates for neoadjuvant chemoradiotherapy followed by surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-26 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Rate of CTCAE acute grade 3 or higher adverse effects possibly attributed to neoadjuvant CRT | Within 90 days of enrollment

SECONDARY OUTCOMES:
Surgical outcomes, including the percentage of patients who undergo a margin-negative (R0) resection and the rate of pathologic complete response (pCR) | Within 30 days following surgery
Rate of postoperative complications | Within 30 days following surgery
Length of hospital stay | Within 30 days following surgery
Rate of CTCAE late grade 3 or higher adverse effects possibly attributed to therapy | 24 months after enrollment
Rate of local-regional recurrence (LRR), progression-free survival (PFS), and overall survival (OS) | 24 months after enrollment
Patient-reported quality of life using LASA-3, Mayo-10, PRO-CTCAE, and FACT-E | 24 months after enrollment
Assessment of early cardiac toxicity after CRT using cardiac MRI | 42 days after completion of CRT

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hallemeier, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials